CLINICAL TRIAL: NCT00934739
Title: Multicentre，A Phase II/III Randomized Study of Adjuvant Anti-Angiogenesis Therapy for Patients of High-Risk Oral Cavity Cancer
Brief Title: A Study of High-Risk Oral Cavity Cancer
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Chang Gung Memorial Hospital (Other); Mackay Memorial Hospital (Other); Changhua Christian Hospital (Other); Sun Yat-sen University (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Veterans General Hospital. (Other); Buddhist Tzu Chi General Hospital (Other); Chi Mei Medical Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1306
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2009-07

CONDITIONS: Oral Cavity Cancer
Keywords: High-Risk Oral Cavity Cancer,; Anti-Angiogenesis
MeSH Terms: conditions — Mouth Neoplasms | interventions — Thalidomide; Celecoxib; Chemotherapy, Adjuvant; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Standard postoperative concurrent chemoradiotherapy
- Thalidomide, Celebrex (Experimental): Adjuvant anti-angiogenesis therapy
  Interventions: Drug: Thalidomide, Celebrex
- Cyclophosphamide, Dexamethasone (Active Comparator): Adjuvant anti-angiogenesis therapy
  Interventions: Drug: Cyclophosphamide, Dexamethasone

INTERVENTIONS:
Drug: Thalidomide, Celebrex — Immediately after operation starts thalidomide (50) 4# per day and celecoxib (Celebrex)(200) 2# bid for three weeks, in addition to standard postoperative concurrent chemoradiotherapy
  Other Names: Adjuvant Therapy
  Arms: Thalidomide, Celebrex
Drug: Cyclophosphamide, Dexamethasone — Immediately after operation starts cyclophosphamide (50) 1# per day and dexamethasone (0.5) 2# qd for three weeks, in addition to standard postoperative concurrent chemoradiotherapy
  Arms: Cyclophosphamide, Dexamethasone

SUMMARY:
Objectives:

1. To study the effect of anti-angiogenesis therapy on reducing the recurrence of high-risk oral cavity cancer patients after curative local treatment.
2. To study the toxicity and compliance of post-operative anti-angiogenesis therapy

Study design:

This is a multi-center randomized controlled phase II/III two-stage study.

Study endpoints:

The primary endpoint is the tumor-free survival (primary and second primary malignancies) and the primary analysis is to compare the tumor-free survival between groups.

DETAILED DESCRIPTION:
Type and number of patients:

Patients with resectable oral cancer of clinical stage N2, 3 or skin-involved T4 will be enrolled.

Sample size at the first stage is 64 patients per group and the total sample size at the end of the second stage is 192 patients per group, assuming that the accrual rate/hazard rate = 1.33, an α=0.05 and power of 0.8 (Hypotheses: H0:θ ≦ 1.0 and Ha: θ ≧ 1.33)

Treatment schedule:

Group A：standard postoperative concurrent chemoradiotherapy.

Group B：Immediately after operation starts thalidomide (50) 4# per day and celecoxib (200) 2# bid for three weeks, in addition to standard postoperative concurrent chemoradiotherapy.

Group C：Immediately after operation starts cyclophosphamide (50) 1# per day and dexamethasone (0.5) 2# qd for three weeks, in addition to standard postoperative concurrent chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proved oral cavity squamous cell carcinoma (buccal and mobile tongue).
2. Clinical stage T4a with skin involvement or resectable N2-3 by UICC/AJCC 1997 staging system.(24)
3. Curative-intent operation feasible and arranged.
4. Eastern Cooperative Oncology Group performance status ≦ 1.
5. A leukocyte count ≧3750/μL, Hb ≧10 g/dL, and a platelet count ≧100,000/μL.
6. A serum bilirubin level < 1.5 UNL (upper normal limit), serum creatinine level < 1.5 UNL or creatinine clearance > 60 mL/min.
7. Age less than 70 years old
8. Informed consent signed.

Exclusion Criteria:

1. Evidence of distant metastatic.
2. Presence of another malignancy other than treated squamous/basal cell carcinoma of the skin.
3. Presence of uncontrolled hypertension, poorly controlled heart failure.
4. Presence of active infection.
5. Patients who have been or are being treated with chemotherapy, radiotherapy, immunotherapy, or other experimental therapies.
6. Women who test positive for pregnancy. Note: Patients received neck lymph node biopsy will be eligible and the stage will be given according to the preoperative status.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the tumor-free survival that is defined as the duration between the dates of operation and the date of disease recurrence. | 7 years

SECONDARY OUTCOMES:
Physical examinations, lab abnormality and other toxicities graded by the NCI Common Toxicity Criteria will be examined to evaluate safety profiles of the study treatments. | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-Long Hong, MD, PhD., Principal Investigator — Department of Oncology, National Taiwan University Hospital